CLINICAL TRIAL: NCT02427373
Title: A Parallel Bioavailability Study of Fish Oil-Ethyl Ester Versus Fish Oil-Triglyceride Versus Krill Oil
Acronym: KOMPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2013-10701
Record Dates: First submitted 2015-04-20; First posted 2015-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Healthy Adults
Keywords: bioavailability; fish oil; krill oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- fish oil ethyl ester (Active Comparator): 1.3g/d dose of DHA+EPA in fish oil EE (6 capsules) administered for 4 weeks
  Interventions: Dietary Supplement: fish oil ethyl ester
- fish oil triglyceride (Active Comparator): 1.3g/d dose of DHA+EPA in fish oil TG (6 capsules) administered for 4 weeks
  Interventions: Dietary Supplement: fish oil triglyceride
- krill oil (Active Comparator): 1.3g/d dose of DHA+EPA in krill oil (6 capsules) administered for 4 weeks
  Interventions: Dietary Supplement: krill oil

INTERVENTIONS:
Dietary Supplement: fish oil ethyl ester
  Arms: fish oil ethyl ester
Dietary Supplement: fish oil triglyceride
  Arms: fish oil triglyceride
Dietary Supplement: krill oil
  Arms: krill oil

SUMMARY:
A multiple-dose, double-blind, randomized, four-week, three-treatment, parallel study in which 66 healthy adult subjects will receive 6 capsules/d, administered as a dose of 1.3 g/d eicosapentaenoic acid (EPA)+docosahexaenoic acid (DHA) in fish oil ethyl ester (EE), or fish oil triglyceride (TG) or krill oil for a total of 4 weeks. The objective of the study is to compare the oral bioavailability of EPA+DHA in total plasma across the three formulations at the end of the 4 week study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy,
* adult female who is neither pregnant nor breastfeeding, or
* a healthy, adult male
* with a body mass index (BMI) between 18 and 30 kg/m2 (inclusive), and
* with a minimum weight of 50 kg (110 lbs).

Exclusion Criteria:

* history or presence of diabetes, high triglycerides (≥240 mg/dL), or high cholesterol (≥240 mg/dL);
* clinically significant abnormal finding on the physical exam, medical history, vital signs, or clinical laboratory results at screening;
* history or presence of allergic response to omega-3-fatty acids or sensitivity or allergy to fish or shellfish;
* history of coagulation disorder or current anticoagulation therapy;
* has used any nutritional supplements, omega-3 supplements, fish oil, chia, krill oil, flaxseed or foods supplemented with omega-3s within 3 months prior to the first dose of study medication;
* has used any prescription medication, except hormonal contraceptive or hormonal replacement therapy, within 14 days prior to the first dose of study medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Comparison of total plasma DHA+EPA levels across 3 treatment groups | 4 weeks

SECONDARY OUTCOMES:
Comparison of RBC DHA+EPA levels across 3 treatment groups | 4 weeks
pharmacokinetic parameter: AUC to 672hr | 4 weeks
pharmacokinetic parameter: AUC to 336hr | 2 weeks
pharmacokinetic parameter: Cmax | 4 weeks
pharmacokinetic parameter: Tmax | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Smeberg, MD, Principal Investigator — Worldwide Clinical Trials

REFERENCES:
- [Derived] Yurko-Mauro K, Kralovec J, Bailey-Hall E, Smeberg V, Stark JG, Salem N Jr. Similar eicosapentaenoic acid and docosahexaenoic acid plasma levels achieved with fish oil or krill oil in a randomized double-blind four-week bioavailability study. Lipids Health Dis. 2015 Sep 2;14:99. doi: 10.1186/s12944-015-0109-z. PMID 26328782